CLINICAL TRIAL: NCT03188094
Title: Integrated Community-Clinical Linkage Model to Promote Weight Loss Among South Asians With Pre-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 17-00693; 1R01DK110048 (NIH)
Record Dates: First submitted 2017-06-06; First posted 2017-06-15 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pre Diabetes; Weight Loss
MeSH Terms: conditions — Glucose Intolerance; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert + CHW-Led Coaching (Experimental): Participants will receive an alert and registry-driven CHW-led coaching during either the first or second round.
  Interventions: Behavioral: CHW-Led Health Coaching; Other: EHR Alerts
- Usual Care - Wait-List Control (No Intervention): All participants waitlisted during the first round will be randomized to the control group. Control group participants will be offered the full CHW group education sessions during the second round. The control participants will receive usual care during the first round.

INTERVENTIONS:
Behavioral: CHW-Led Health Coaching — The CHW intervention includes a protocol that consists of 5 monthly 90-minute group health education sessions, providing the tools and strategies to prevent diabetes.
  Arms: Alert + CHW-Led Coaching
Other: EHR Alerts — Primary care providers (PCP) treating patients in the intervention group will receive embedded EHR alerts to increase screening and identification of South Asian patients at-risk for T2DM with BMI >23 kg/m2 and registries to track outcomes.
  Arms: Alert + CHW-Led Coaching

SUMMARY:
The proposed study will inform efforts to prevent diabetes and promote weight loss in a high-risk population and generate a reproducible, scalable, and sustainable model for use with other insurer groups and clinical settings that work in immigrant populations with a high burden of chronic disease.

DETAILED DESCRIPTION:
The study "Integrated Community-Clinical Linkage Model to Promote Weight Loss among South Asians with Pre-Diabetes" aims to test the effectiveness and assess the implementation process of an integrated intervention to support weight loss for South Asian patients at-risk for type-2 diabetes mellitus (T2DM) in primary care settings. The integrated intervention involves:

1. An electronic health record (EHR) intervention for primary care providers (PCPs) utilizing embedded alerts to increase screening and identification of South Asian patients at-risk for T2DM with BMI >23 kg/m2 and registries to track outcomes: and
2. Registry-driven community health worker (CHW)-led health coaching for patients. Using a stepped-wedge design, we will implement the study in 25 New York City PCP sites enrolling 2,840 South Asian patients at- risk for T2DM.
3. Provider Surveys (n=40) to capture data on satisfaction with workflow before and after intervention, information sources for EHR-CHW initiatives before and after intervention, acceptability of and satisfaction with the integrated EHR-CHW intervention, and barriers and facilitators of point-of-care use of the tools.
4. Key Informant Interviews (n=35) with physician champions at each site and/or administrator of each site, Health first representatives, and CHWs. At baseline, the interviews will be incorporated into the workflow analysis to assess current satisfaction and usage of EHR and health coaching. At follow-up, the interviews will assess barriers and facilitators to the implementation and adoption process of the integrated EHR-CHW intervention, fidelity to the interventions, and to solicit recommendations for the replication and scalability of the intervention to other sites and insurer organizations.

ELIGIBILITY:
Inclusion Criteria:

* self identify as South Asian;
* are at least 21 years of age and younger than age 75,
* had an appointment with a physician or mid-level clinician for routine non-emergent primary care in the last 12 months;
* have a BMI of >23; and
* have incident pre-diabetes as determined by HbA1c test (last A1c test date in the last 12 months).

Exclusion Criteria:

* Patients under the age of 21 and older than 75 will be excluded.
* Individuals with a diagnosis of diabetes or pre-diabetes during the 12 months prior to intervention implementation will be excluded.
* Pregnant women and all visits with an obstetrician gynecologist are excluded.
* No children or vulnerable subjects will be enrolled in this study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- [Derived] Gupta A, Wyatt LC, Mammen S, Zanowiak JM, Lim S, Islam NS, Kumar R, Beane S, Gold HT. Cost analysis of implementing a community health worker-led weight reduction randomized-controlled trial among prediabetic south asian patients at primary care sites in NYC. Implement Sci. 2025 Jun 2;20(1):26. doi: 10.1186/s13012-025-01439-2. PMID 40457309
- [Derived] Hu L, Wyatt LC, Mohsin F, Lim S, Zanowiak J, Mammen S, Hussain S, Ali SH, Onakomaiya D, Belli HM, Aifah A, Islam NS. Characterizing Technology Use and Preferences for Health Communication in South Asian Immigrants With Prediabetes or Diabetes: Cross-Sectional Descriptive Study. JMIR Form Res. 2024 Apr 26;8:e52687. doi: 10.2196/52687. PMID 38669062
- [Derived] Lim S, Wyatt LC, Mammen S, Zanowiak JM, Mohaimin S, Goldfeld KS, Shelley D, Gold HT, Islam NS. The DREAM Initiative: study protocol for a randomized controlled trial testing an integrated electronic health record and community health worker intervention to promote weight loss among South Asian patients at risk for diabetes. Trials. 2019 Nov 21;20(1):635. doi: 10.1186/s13063-019-3711-y. PMID 31752964

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Primary care providers (PCPs) were not considered enrolled as participants in this study.
Units Other Than Participants: Clinics
Groups:
- Waive 1 (10/2018-12/2019) Round 1 Jan-Jun 2019, Round 2 July-Dec 2019: All participants waitlisted during the Waive 1- Round 1 were randomized to the Waive 1 Wait-List Control group.
  During the first round (Jan-Jun 2019), participants received standard of care. During the second round (July-Dec 2019), all control participants were offered the full CHW group education sessions, though not for research purposes.
  Participants randomized to receive the intervention in Waive 1 received the intervention from Jan-Jun 2019 for Round 1; Round 2 participants received the intervention from July-Dec 2019.
- Waive 2 (10/2019-12/2020) Round 1 Jan-Jun 2020, Round 2 July-Dec 2020: All participants waitlisted during the Waive 2 - Round 1 were randomized to the Waive 2 Wait-List Control group.
  During the first round (Jan-Jun 2020), participants received standard of care. During the second round (July-Dec 2020), all control participants were offered the full CHW group education sessions, though not for research purposes.
  Participants randomized to receive the intervention in Waive 2 received the intervention from Jan-Jun 2020 for Round 1; Round 2 participants received the intervention from July-Dec 2020.
- Waive 3 (10/2020-12/2021) Round 1 Jan-Jun 2021, Round 2 July-Dec 2021: All participants waitlisted during the Waive 3 - Round 1 were randomized to the Waive 3 Wait-List Control group.
  During the first round (Jan-Jun 2021), participants received standard of care. During the second round (July-Dec 2021), all control participants were offered the full CHW group education sessions, though not for research purposes.
  Participants randomized to receive the intervention in Waive 3 received the intervention from Jan-Jun 2021 for Round 1; Round 2 participants received the intervention from July-Dec 2021.
Period: Overall Study
Arm/Group | Waive 1 (10/2018-12/2019) Round 1 Jan-Jun 2019, Round 2 July-Dec 2019 | Waive 2 (10/2019-12/2020) Round 1 Jan-Jun 2020, Round 2 July-Dec 2020 | Waive 3 (10/2020-12/2021) Round 1 Jan-Jun 2021, Round 2 July-Dec 2021
Started | 333; 7 Clinics | 294; 7 Clinics | 347; 5 Clinics
Participants Started Wait-List Control Round 1, CHW Round 2 | 164; 7 Clinics | 147; 7 Clinics | 165; 5 Clinics
Participants Completed Wait-List Control Round 1, CHW Round 2 | 164; 7 Clinics | 147; 7 Clinics | 165; 5 Clinics
Participants Started CHW Round 1, CHW Round 2 | 169; 7 Clinics | 147; 7 Clinics | 182; 5 Clinics
Participants Completed CHW Round 1, CHW Round 2 | 164; 7 Clinics | 147; 7 Clinics | 165; 5 Clinics
Completed | 328; 7 Clinics | 294; 7 Clinics | 330; 5 Clinics
Not Completed | 5; 0 Clinics | 0; 0 Clinics | 17; 0 Clinics
Not completed — Screen failure | 1 | 0 | 0
Not completed — Pregnancy | 3 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care - Wait-List Control | Alert + CHW-Led Coaching | Total
Number analyzed (Participants) | 476 | 476 | 952
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.2) | 48.2 (11.2) | 48.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 274 | 548
  Male | 202 | 202 | 404
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 476 | 476 | 952
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 476 | 476 | 952
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 476 | 476 | 952

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Lost at Least 5% of Body Weight Between Baseline and Month 6
Description: Weight measured at baseline and 6 month survey via study scale.
Time Frame: Baseline, Month 6
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care - Wait-List Control | Alert + CHW-Led Coaching
Number analyzed (Participants) | 210 | 457
Percentage of participants | 11 | 19

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care - Wait-List Control | Alert + CHW-Led Coaching
All-Cause Mortality (participants affected / at risk) | 0/476 | 0/498
Serious Adverse Events (participants affected / at risk) | 0/476 | 0/498
Other Adverse Events (participants affected / at risk) | 0/476 | 0/498

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03188094/Prot_SAP_000.pdf